CLINICAL TRIAL: NCT00677859
Title: A Phase I, Multicenter, Dose-Escalation Trial Evaluating Maximum-Tolerated Dose of Single and Repeated Administration of Allogeneic MultiStem® in Patients With Acute Leukemia, Chronic Myeloid Leukemia, or Myelodysplasia
Brief Title: Safety Study of MultiStem® in Patients With Acute Leukemia, Chronic Myeloid Leukemia, or Myelodysplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Healios K.K. (Industry)
Collaborators: Cato Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GVHD-2007-001
Record Dates: First submitted 2008-05-14; First posted 2008-05-15 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Hematologic Malignancies
Keywords: Leukemia; Graft vs. Host Disease; Hematopoietic Stem Cell Transplant; Bone Marrow Transplant; Myelodysplasia
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Graft vs Host Disease; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single dose Arm (Experimental): There will be six cohorts of three patients each. Three escalating doses of MultiStem will be evaluated.
  Interventions: Biological: MultiStem®
- Repeat Dose Arm (Experimental): There will be six cohorts of three patients each. Four dosing regimens will be evaluated,varying doses at three times weekly or five times weekly.
  Interventions: Biological: MultiStem®

INTERVENTIONS:
Biological: MultiStem® — Patients will receive a single IV infusion of MultiStem® 2 days after HSCT.
  Arms: Single dose Arm
Biological: MultiStem® — Patients will receive either 3 weekly IV infusions or 5 weekly infusions of MultiStem®
  Arms: Repeat Dose Arm

SUMMARY:
The purpose of this study is to determine if MultiStem® can safely be given to patients with acute leukemia, chronic myeloid leukemia, or myelodysplasia after they have received hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Graft-vs.-Host Disease (GVHD) is one of the major limitations of allogeneic hematopoietic stem cell transplants (HSCT). This complication is major cause of morbidity and mortality and is thought to be initiated by activation of donor T-cells through recognition of "foreign" cells resident in the transplant recipient. Acute GVHD is associated with damage to the liver, skin, gastrointestinal tract and mucosa. Moderate to severe GVHD Grades II-IV occurs in 30-50% of matched related HSCTs and 50-70% of unrelated donor recipients. Severe GHVD requires intense immunosuppression involving steroids and additional agents to get it under control, and patients may develop severe infections as a result of such immunosuppression. An agent or cell therapy that could reduce the incidence and/or severity of GVHD without increasing relapse or infectious risk in HSCT patients would provide substantial benefits.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged 18-65 years of age
* Diagnosis of acute myeloid or lymphoblastic leukemia (second or subsequent remission, if not in remission, then <20% bone marrow blasts), chronic myelogenous leukemia resistant to or intolerant of tyrosine kinase inhibitor therapy (accelerated phase, first chronic phase with TKI resistance, or second chronic phase), or myelodysplastic syndrome (intermediate/high or high risk by International Prognostic Scoring System (IPSS), lower risk by IPSS with patient having progressed after prior therapy. Complete remission is defined as the absence of blasts in the peripheral circulation at the time of enrollment and <5% blasts in the marrow within 28 days of enrollment.
* Life expectancy of at least 100 days
* Patients scheduled for allogeneic bone marrow transplant or peripheral blood stem cell transplant (PBST) procedure
* Family-related or unrelated donors
* HLA matching should either be matched related or matched unrelated donors, 6/6 match or 5/6 single allelic mismatch, with provision that the DRB1 is molecularly matched
* Performance status (ECOG ≤2)
* Signed informed consent

Exclusion Criteria:

* Active infection
* Known allergies to bovine or porcine products
* Renal function: Serum creatinine >2 mg/dL or creatinine clearance ≤50 mL/min
* Hepatic function: Screening ALT or AST ≥3x than the upper limit of normal for the laboratory OR total bilirubin ≥2.0 mg/dL (Exception: acceptable if patient is identified with pre-existing condition e.g., Gilbert's disease that will contribute to baseline elevations of bilirubin)
* Pulmonary function: FEV1, FVC, DLCO ≤50% predicted
* Cardiac function: left ventricular ejection fraction ≤50%
* Patient received an investigational agent within 30 days prior to transplant
* The patient is pregnant, has a positive serum BhCG, or is lactating
* Patient on corticosteroids at a dose >0.25 mg/kg/day
* Planned non-myeloablative transplant
* Planned cord blood transplant
* Prior allogeneic myeloablative HSCT
* HIV seropositive, HTLV seropositive, hepatitis B or C seropositive, varicella virus active infection, or syphilis active infection
* Other serious medical or psychiatric illness that, in the investigator's opinion, would not permit the patient to be managed according to the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-07; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 30 days

SECONDARY OUTCOMES:
incidence of grade III/IV GVHD | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Maziarz, MD, Principal Investigator — Oregon Health and Science University; Steven Devine, MD, Principal Investigator — Ohio State University; Hillard Lazarus, MD, Principal Investigator — Case Western Reserve University
Locations (6):
- United States (5):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Oregon State University Medical Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Transplant Institute, San Antonio, Texas
- UZ Leuven, Leuven, Belgium